CLINICAL TRIAL: NCT03332108
Title: Novel Approach to Improving Lactation Support Using Mobile Health Technology
Brief Title: Novel Approach To Improving Lactation Support With Mobile Health Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other); Washington University Institute of Clinical and Translational Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201705027
Record Dates: First submitted 2017-09-13; First posted 2017-11-06 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Breastfeeding; Feeding Behavior
Keywords: mobile health (mHealth); electronic health (eHealth); breastfeeding; infant nutrition; text messaging intervention
MeSH Terms: conditions — Breast Feeding; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Those allocated to the intervention arm will be enrolled in the mHealth intervention (EpxBreastfeeding) for six months, and will also be asked about breastfeeding status at their six-week postpartum follow up visit (standard of care) as well as during phone interviews at three and six months postpartum.
  Interventions: Other: EpxBreastfeeding; Other: Baby book survey
- Control (Other): Those in the control arm will be asked about breastfeeding status (exclusive, supplementing, or formula only) at their six-week postpartum follow up visit (standard of care) as well as during phone interviews at three and six months postpartum.
  Interventions: Other: Baby book survey

INTERVENTIONS:
Other: EpxBreastfeeding — We developed an algorithm using the Epharmix platform, an automated toll-free phone and text message-based system that can programmatically query patients via their personal phones and subsequently collect response data, allowing clinically-relevant responses to trigger alerts to designated healthcare providers. The intervention for breastfeeding, hereafter referred to as EpxBreastfeeding, was built using significant clinical and patient input to only ask the most clinically-relevant questions for breastfeeding in a multiple-choice manner, such as "In the past [x] days, have you fed your baby 1) breast milk only, 2) breast milk and formula or 3) formula only?". These communications elicit patient-reports of breastfeeding at intervals of interest for the provider, which is, on average, every 2 days in the first three weeks postpartum and every 5 days subsequently. All data is filtered by clinician-designed algorithms to stratify patients into categories.
  Arms: Intervention
Other: Baby book survey — We developed a "baby book" template that will be given to mothers allowing them to make note of dates related to their child's development during the first year. Examples include: When was baby's first appointment with his/her pediatrician? When did you add formula into baby's feeding? When did you start feeding baby only formula? When did you introduce solid food into baby's diet? When did baby first smile? When did you start reading to baby? What was the first book you read to baby? Whe

SUMMARY:
This is a randomized trial of use of a mobile health tool (EpxBreastfeeding) aimed at improving breastfeeding adherence and duration among recent mothers who self identify as motivated to breastfeed. As a result of text communication and expedited coaching through common breastfeeding challenges, the investigators expect more mothers in the study arm will continue breastfeeding through the first 6 months after giving birth.

DETAILED DESCRIPTION:
Immediately following delivery, mothers are given the task of learning to care for a newborn, coping with rapid hormone changes, and in many cases, learning to breastfeed, all with minimal contact with their obstetric provider. Traditionally, women are not seen by their obstetrician until 6 weeks postpartum, increasing the likelihood that they will switch to formula feeding despite a clear antenatal intent to breastfeed.

Data suggests that exclusive breastfeeding for the first six months of life is associated with lower rates of respiratory and ear infections in babies with fewer required hospitalizations, due to the protective effect of maternal antibodies in breast milk. Fewer children go on to develop asthma and allergies. Additionally, adolescents who were breastfed demonstrate higher intelligence quotient (IQ) averages that their peers who were not. The benefits of breastfeeding for mothers include healthy weight loss and protection against ovarian and breast cancer, as well as psychological wellness through maternal-infant bonding. The World Health Organization (WHO) has published extensive data to support recommendations for exclusive breastfeeding in the first 6-month period. Exclusive breastfeeding is defined as the infant's only source of nutrition being human breast milk (along with vitamins, minerals, and medications). While the WHO and the American Congress of Obstetricians and Gynecologists (ACOG) recommend 6 months of exclusive breastfeeding, data published by the Centers for Disease Control (CDC) in 2016 show that only 81.1% of mothers ever try breastfeeding, only 44.4% exclusively breastfeed through 3 months, and only 22.3% exclusively breastfeed over 6 months. In Missouri, the CDC's report card data shows that 85.4% of mothers ever breastfed, and rates of exclusive breastfeeding were 49.7% and 24.7% at 3 and 6 months respectively. At the investigators' local hospital, a recent chart review as part of the Barnes Jewish Hospital's Baby Friendly designation process demonstrated that only 45% of mothers who received prenatal care at the Center for Advanced Medicine (CAM) or the Center for Outpatient Health (COH) were exclusively breastfeeding at 6 weeks postpartum (unpublished data). In order to reach the Healthy People 2020 goals of 42.6% breastfeeding at 3 months and 60.6% at 6 months, it is important to identify modifiable barriers to optimal breastfeeding practices and create innovative solutions to address them.

One of these barriers is access to lactation support. Mothers frequently have difficulty becoming familiar with the process of breastfeeding during the immediate postpartum period. "Difficulty latching" or "inadequate milk production" are the most common causes of concern, driving mothers to supplement with or switch to milk formula products. Once efforts to breastfeed cease, mammary milk production slows and cannot be restarted. Mothers who have started formula feeds at time of discharge from the hospital are five times more likely to stop breastfeeding completely in the first week. The ACOG strongly supports breastfeeding, recognizing it as a public health priority, and has promoted the implementation of clinical resources in hospital systems nationwide. Many hospitals employ dedicated professionals trained in breastfeeding (lactation consultants and obstetric and postpartum nurses trained specifically in lactation support) to counsel and assist mothers, and the use of lactation consultants has been shown to significantly increase breastfeeding rates. Unfortunately, trends show that after mothers and infants are discharged from the hospital, they lose connection with these providers. The lack of support is one of many factors that may lead to cessation of exclusive breastfeeding.

In typical postpartum practice, patients return to their obstetrics provider for a visit at 6 weeks. This is inadequate for addressing breastfeeding concerns, as it occurs too late to promote a return to a breastfeeding. Proactive outreach in busy obstetrics practices is expensive, time-consuming and inefficient due to challenges with identifying and targeting resources to mothers who are most in need of a help achieving their breastfeeding goals. Postpartum visits are, by default, included in a patient's global obstetric package and providers are in many cases unable to bill separately for lactation support visits, which can make it harder for mothers and providers to address issues earlier postpartum. Ideally, an approach to improving patient/provider communication in the 2 postpartum weeks when most breastfeeding challenges arise would provide support out of the office setting, with follow up through 6 months. The system must ideally be low cost, low tech, and efficient enough to be implemented widely. Short message service (SMS) texting interventions mark a novel entry point to the healthcare field and enable targeting to patients across the socioeconomic spectrum. Every cell phone is equipped for SMS texting. This form of communication also allows the patient to respond to prompt messages, thereby reducing the burden on patients to initiate communication.

Breastfeeding improves maternal and infant health. Most expert bodies recommend at least 6 months of exclusive breastfeeding. Unfortunately, breastfeeding can be difficult to start and sustain due to a variety of mostly treatable factors; many mothers are currently left to navigate these difficulties on their own. The investigators hypothesize that close and individualized assistance will increase the rates of exclusive breastfeeding. To achieve this, a novel, automated, two-way text messaging platform has been developed. This system offers encouragement and education but perhaps more importantly, it collects and categorizes feedback from each mother to identify those that may benefit from personalized follow-up by a trained professional. This system was developed by a team of students and healthcare professionals. The investigators propose implementing it in obstetrics clinics at BJH, and will study its impact through quantitative measures and feedback. If successful, this proposal will create a scalable technological solution to improve breastfeeding adherence.

Hypothesis:

An automated bidirectional communication tool (EpxBreastfeeding) to monitor nursing status and assess for common problems related to breastfeeding will improve provider awareness and expedite personal follow-up with patients identified as at risk of stopping breastfeeding, and will improve breastfeeding adherence over time compared to controls.

Specific Aims:

1. Determine if exclusive breastfeeding duration can be improved by using an automated bidirectional communication tool compared to standard of care through six months postpartum.
2. Compare time-to-event incidence reporting and subsequent provider response time to duration of breastfeeding status (intervention cohort only).
3. Collect subjective data from mothers receiving the intervention, as well as ancillary professionals who are designated for notification and follow-up to consider the feasibility and acceptance of an automated bidirectional mHealth lactation support intervention in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 to 40 years
* Singleton birth (e.g. no twins or triplets)
* Prenatal intention to breastfeed
* Have a mobile phone capable of receiving SMS text messages and phone calls
* Know how to send a text message
* ≥4th grade literacy level

Exclusion Criteria:

* Non-fluent in English
* Known fetal anomaly
* Infant delivery <37 weeks
* >3 days in neonatal intensive care unit (NICU)
* Medical history: pre-pregnancy BMI >50, history of thyroid disorders, failed one hour and three hour glucola test or if they ever needed oral hypoglycemic, hypertension (HTN) before/during pregnancy, postpartum hemorrhage
* Medically contraindicated for breastfeeding (provider's judgment)
* Women who will breastfeed but not from their own breast (e.g. buy breast milk on the Internet/milk bank)
* Women who are hesitant about answering a series of text messages regularly
* Women who are unable to be contacted by SMS text message or are unwilling to provide their contact number
* Women with neurologic, anatomic, or cognitive disorders that are unable to consent and/or answer text messages

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women having given birth with the intention to breastfeed
Enrollment: 218 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding duration | Six months
  The primary outcome is the length of time mothers exclusively breastfeed (i.e. continuous length of time for which mothers only give breast milk).

SECONDARY OUTCOMES:
Time to transition feeding status | Six months
  Time to transition from exclusive breastfeeding to partial breastfeeding (supplementing breast milk with formula) as well as supplemental nursing only.
Time to event | Six months
  Time to reported problems with: latching, concern regarding deficiency in milk production, concern for inadequate child's weight gain

OTHER OUTCOMES:
Time from event to provider intervention | Six months
  Time from reported lactation/nursing problem to provider intervention.
Time to nursing status change | Six months
  Time from provider intervention to change in nursing status (exploratory analysis of each problem reported)
Engagement | Six months
  Weekly, monthly, and gross response rate to text messages
Patient Satisfaction with Provider, Service and Survey | Six months
  Patient satisfaction with provider, communication with provider, frequency of messages, and how likely to recommend the service to a friend measured by automated quality surveys sent each month, with quality ratings of 1-9.
Breastfeeding status at 6 weeks postpartum | Six weeks
  Compare the proportion of mothers exclusively breastfeeding, mixed feeding, and formula feeding at 6 weeks postpartum between control and intervention arms
Breastfeeding status at 3 months postpartum | Three months
  Compare the proportion of mothers exclusively breastfeeding, mixed feeding, and formula feeding at 3 months postpartum between control and intervention arms
Proportion of mothers exclusively breastfeeding at 6 months postpartum | Six months
  Compare the proportion of mother exclusively breastfeeding at 6 months postpartum between control and intervention arms

CONTACTS AND LOCATIONS:
Overall Officials: Camaryn Chrisman Robbins, MD, MPH, Principal Investigator — Associate Professor and Co-Medical Director of Labor and Delivery, Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Hanieh S, Ha TT, Simpson JA, Thuy TT, Khuong NC, Thoang DD, Tran TD, Tuan T, Fisher J, Biggs BA. Exclusive breast feeding in early infancy reduces the risk of inpatient admission for diarrhea and suspected pneumonia in rural Vietnam: a prospective cohort study. BMC Public Health. 2015 Nov 24;15:1166. doi: 10.1186/s12889-015-2431-9. PMID 26602368
- [Background] Horta BL, Loret de Mola C, Victora CG. Breastfeeding and intelligence: a systematic review and meta-analysis. Acta Paediatr. 2015 Dec;104(467):14-9. doi: 10.1111/apa.13139. PMID 26211556
- [Background] Horta BL, Loret de Mola C, Victora CG. Long-term consequences of breastfeeding on cholesterol, obesity, systolic blood pressure and type 2 diabetes: a systematic review and meta-analysis. Acta Paediatr. 2015 Dec;104(467):30-7. doi: 10.1111/apa.13133. PMID 26192560
- [Background] Patel S, Patel S. The Effectiveness of Lactation Consultants and Lactation Counselors on Breastfeeding Outcomes. J Hum Lact. 2016 Aug;32(3):530-41. doi: 10.1177/0890334415618668. Epub 2015 Dec 7. PMID 26644419
- [Background] Tahir NM, Al-Sadat N. Does telephone lactation counselling improve breastfeeding practices? A randomised controlled trial. Int J Nurs Stud. 2013 Jan;50(1):16-25. doi: 10.1016/j.ijnurstu.2012.09.006. Epub 2012 Oct 17. PMID 23084438
- [Background] Chung M, Ip S, Yu W, Raman G, Trikalinos T, DeVine D, Lau J. Interventions in Primary Care to Promote Breastfeeding: A Systematic Review [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Oct. Report No.: 09-05126-EF-1. Available from http://www.ncbi.nlm.nih.gov/books/NBK35168/ PMID 20722164
- [Background] Fiscella K, Franks P, Gold MR, Clancy CM. Inequality in quality: addressing socioeconomic, racial, and ethnic disparities in health care. JAMA. 2000 May 17;283(19):2579-84. doi: 10.1001/jama.283.19.2579. PMID 10815125
- [Background] Lua PL, Neni WS. A randomised controlled trial of an SMS-based mobile epilepsy education system. J Telemed Telecare. 2013 Jan;19(1):23-8. doi: 10.1177/1357633X12473920. Epub 2013 Feb 6. PMID 23390210
- [Background] Jerant A, Sohler N, Fiscella K, Franks B, Franks P. Tailored interactive multimedia computer programs to reduce health disparities: opportunities and challenges. Patient Educ Couns. 2011 Nov;85(2):323-30. doi: 10.1016/j.pec.2010.11.012. Epub 2010 Dec 13. PMID 21146950
- [Background] Moniz MH, Meyn LA, Beigi RH. Text Messaging to Improve Preventive Health Attitudes and Behaviors During Pregnancy: A Prospective Cohort Analysis. J Reprod Med. 2015 Sep-Oct;60(9-10):378-82. PMID 26592061
- [Background] McFadden A, Gavine A, Renfrew MJ, Wade A, Buchanan P, Taylor JL, Veitch E, Rennie AM, Crowther SA, Neiman S, MacGillivray S. Support for healthy breastfeeding mothers with healthy term babies. Cochrane Database Syst Rev. 2017 Feb 28;2(2):CD001141. doi: 10.1002/14651858.CD001141.pub5. PMID 28244064
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- See also: Clinical guidelines: breastfeeding. American College of Obstetrics and Gynecologists — http://www.acog.org/About-ACOG/ACOG-Departments/Breastfeeding